CLINICAL TRIAL: NCT01767974
Title: Comparison of Sequencing and PNA Clamping of EGFR Gene in Patients With Non-Small Cell Type Lung Cancer
Acronym: SPACE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chonnam National University Hospital (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Young-Chul Kim, Professor, Chonnam National University Hospital
Other Study IDs: ISSIRES0066
Record Dates: First submitted 2013-01-11; First posted 2013-01-15 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2013-01

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-Small Cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA from lung cancer tumor tissue obtained by bronchoscopy, needle biopsy or surgical resection
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Non-Small Cell Lung Cancer: Locally advanced stage IIIB or IV (metastatic) or Relapsed Non-Small Cell Lung Cancer

SUMMARY:
Using DNA acquired from tumor tissue, sequencing and PNA-clamping for EGFR gene will be performed. The detection rates of EGFR mutation will be compared using paired samples.

DETAILED DESCRIPTION:
Single arm, open label, prospective, observational study of gefitinib treatment for locally advanced (stage IIIB) or IV (metastatic) or relapsed NSCLC patients.

Using DNA acquired from tumor tissue, sequencing and PNA-clamping for EGFR gene will be performed. The detection rates of EGFR mutation will be compared using paired samples.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced stage IIIB not suitable for curative therapy or stage IV (metastatic) disease or relapsed NSCLC
* ECOG Performance status 0~2.
* Written Informed Consent
* Female or male patients aged 18 years or over, eligible for treatment for NSCLC

Exclusion Criteria:

* Previous exposure to EGFR-TKI
* Concomitant use of other anti-cancer drugs with EGFR-TKI
* Patients without available Tumor DNA
* As judged by the investigator, any evidence of severe or uncontrolled systemic disease (e.g. unstable or uncompensated respiratory, cardiac, hepatic, or renal disease)
* Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the subject to participate in the study
* Pregnancy or breast-feeding women (women of child¬bearing potential). Women of childbearing potential must practice acceptable methods of birth control to prevent pregnancy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Locally advanced stage IIIB or IV (metastatic) or Relapsed Non-Small Cell Lung Cancer
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-12 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Detection rate of EGFR mutation | two weeks
  To prove higher detection rate of EGFR mutation with PNA clamping compared with sequencing

SECONDARY OUTCOMES:
Verification of PNA positive casese | Two weeks
  To analyze the Sequencing negative/PNA clamping positive group (where sample is available) with another sensitive technique COBAS test

CONTACTS AND LOCATIONS:
Overall Officials: Young-Chul Kim, MD, PhD, Principal Investigator — Chonnam National University Hospital
Locations (1):
- Chonnam National University Hwasun Hospital, Hwasun-Gun, Jeollanam-do, South Korea